CLINICAL TRIAL: NCT00850538
Title: The Role of Bone and Its Measurement in Knee Osteoarthritis
Brief Title: Role of Bone in Knee Osteoarthritis (OA)
Status: Completed | Type: Observational
Sponsor: The New England Baptist Hospital (Other)
Responsible Party: Principal Investigator, David Hunter, PI, The New England Baptist Hospital
Other Study IDs: NEBH 2008-018
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Results first posted 2015-12-04 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-11

CONDITIONS: Osteoarthritis, Knee
Keywords: Bone Marrow Lesion; BML; Arthroplasty; Replacement; Knee; Discarded tissue
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tibial plateau patella fat pad synovial fluid and synovium
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: MRI — 1.5T MRI exam of signal knee with knee coil (estimated time: 35 minutes)
Procedure: Primary Total Knee Replacement — Fluid, bone, and meniscus specimens obtained from total joint replacement will be collected.

SUMMARY:
The purpose of the study is to investigate protein and gene expression among damaged knee tissues. We will perform MRI's on subjects prior to total knee replacement to identify the location of bone marrow lesions. Connective tissues including tendon, ligament, and meniscus specimens normally discarded from total joint replacements will be used for live cell harvest, and protein and gene expression analyses of tissue or cultured cells.

DETAILED DESCRIPTION:
BACKGROUND AND SIGNIFICANCE:

Although the presence of bone marrow lesions (BML) on MRI is strongly associated with osteoarthritis (OA) progression and pain in some studies, the mechanism for this relation and the underlying pathology is not well established. The lack of knowledge on what these lesions constitute hampers their clinical utility both with regards to measurement and targeting for therapeutic intervention.

Our preliminary data has localized specific changes in bone mineralization, remodeling and defects within BML features that are adjacent to the subchondral plate. BMLs appear to be sclerotic compared to unaffected regions; however, the mineral density in these lesions is reduced and may render this area to be mechanically compromised, and thus susceptible to attrition. Limited histological analysis of BMLs reveal thrombi, diffuse fibrinoid necrosis and hyperplasia of blood vessel walls - all indicative of infarction-like pathology.

The aim of this research proposal is to create more specific targets and improve our understanding of the pathology in BMLs.

Specific Aim 1:

- To collect tissue to evaluate protein and gene expression of these tissues and cultured cells.

ELIGIBILITY:
Inclusion Criteria:

* subjects having primary knee replacement surgery with 1 participating surgeon at NEBH (principal investigator)

Exclusion Criteria:

* subjects having a revision knee replacement instead of a primary knee replacement
* contraindications for MRI
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male or female, over age 18, with scheduled primary total knee replacement surgery at NEBH, with no contradindications for MRI
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2008-07; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hunter, MD, Principal Investigator — University of Sydney
Locations (1):
- University of Sydney, Sydney, New South Wales, Australia

REFERENCES:
- [Background] Burr DB. The importance of subchondral bone in the progression of osteoarthritis. J Rheumatol Suppl. 2004 Apr;70:77-80. No abstract available. PMID 15132360
- [Background] Felson DT, Chaisson CE, Hill CL, Totterman SM, Gale ME, Skinner KM, Kazis L, Gale DR. The association of bone marrow lesions with pain in knee osteoarthritis. Ann Intern Med. 2001 Apr 3;134(7):541-9. doi: 10.7326/0003-4819-134-7-200104030-00007. PMID 11281736
- [Background] Felson DT, McLaughlin S, Goggins J, LaValley MP, Gale ME, Totterman S, Li W, Hill C, Gale D. Bone marrow edema and its relation to progression of knee osteoarthritis. Ann Intern Med. 2003 Sep 2;139(5 Pt 1):330-6. doi: 10.7326/0003-4819-139-5_part_1-200309020-00008. PMID 12965941
- [Background] Lo GH, Hunter DJ, Zhang Y, McLennan CE, Lavalley MP, Kiel DP, McLean RR, Genant HK, Guermazi A, Felson DT. Bone marrow lesions in the knee are associated with increased local bone density. Arthritis Rheum. 2005 Sep;52(9):2814-21. doi: 10.1002/art.21290. PMID 16145676
- [Background] Hunter DJ, Zhang Y, Niu J, Goggins J, Amin S, LaValley MP, Guermazi A, Genant H, Gale D, Felson DT. Increase in bone marrow lesions associated with cartilage loss: a longitudinal magnetic resonance imaging study of knee osteoarthritis. Arthritis Rheum. 2006 May;54(5):1529-35. doi: 10.1002/art.21789. PMID 16646037
- [Background] Zanetti M, Bruder E, Romero J, Hodler J. Bone marrow edema pattern in osteoarthritic knees: correlation between MR imaging and histologic findings. Radiology. 2000 Jun;215(3):835-40. doi: 10.1148/radiology.215.3.r00jn05835. PMID 10831707
- [Background] Neuhold A, Hofmann S, Engel A, Leder K, Kramer J, Haller J, Plenk H. Bone marrow edema of the hip: MR findings after core decompression. J Comput Assist Tomogr. 1992 Nov-Dec;16(6):951-5. doi: 10.1097/00004728-199211000-00023. PMID 1430447
- [Background] Plenk H Jr, Hofmann S, Eschberger J, Gstettner M, Kramer J, Schneider W, Engel A. Histomorphology and bone morphometry of the bone marrow edema syndrome of the hip. Clin Orthop Relat Res. 1997 Jan;(334):73-84. PMID 9005898
- [Background] Reinus WR, Fischer KC, Ritter JH. Painful transient tibial edema. Radiology. 1994 Jul;192(1):195-9. doi: 10.1148/radiology.192.1.8208937.
- [Background] Hunter DJ, Lo GH, Gale D, Grainger AJ, Guermazi A, Conaghan PG. The reliability of a new scoring system for knee osteoarthritis MRI and the validity of bone marrow lesion assessment: BLOKS (Boston Leeds Osteoarthritis Knee Score). Ann Rheum Dis. 2008 Feb;67(2):206-11. doi: 10.1136/ard.2006.066183. Epub 2007 May 1. PMID 17472995
- [Background] Kornaat PR, Bloem JL, Ceulemans RY, Riyazi N, Rosendaal FR, Nelissen RG, Carter WO, Hellio Le Graverand MP, Kloppenburg M. Osteoarthritis of the knee: association between clinical features and MR imaging findings. Radiology. 2006 Jun;239(3):811-7. doi: 10.1148/radiol.2393050253. PMID 16714463
- [Background] Hayes CW, Jamadar DA, Welch GW, Jannausch ML, Lachance LL, Capul DC, Sowers MR. Osteoarthritis of the knee: comparison of MR imaging findings with radiographic severity measurements and pain in middle-aged women. Radiology. 2005 Dec;237(3):998-1007. doi: 10.1148/radiol.2373041989. Epub 2005 Oct 26. PMID 16251398
- [Background] Simkin PA. Bone pain and pressure in osteoarthritic joints. Novartis Found Symp. 2004;260:179-86; discussion 186-90, 277-9. PMID 15283450
- [Background] Mach DB, Rogers SD, Sabino MC, Luger NM, Schwei MJ, Pomonis JD, Keyser CP, Clohisy DR, Adams DJ, O'Leary P, Mantyh PW. Origins of skeletal pain: sensory and sympathetic innervation of the mouse femur. Neuroscience. 2002;113(1):155-66. doi: 10.1016/s0306-4522(02)00165-3. PMID 12123694
- [Background] Hukkanen M, Konttinen YT, Rees RG, Gibson SJ, Santavirta S, Polak JM. Innervation of bone from healthy and arthritic rats by substance P and calcitonin gene related peptide containing sensory fibers. J Rheumatol. 1992 Aug;19(8):1252-9. PMID 1383542
- [Background] Hunter DJ, Gerstenfeld L, Bishop G, Davis AD, Mason ZD, Einhorn TA, Maciewicz RA, Newham P, Foster M, Jackson S, Morgan EF. Bone marrow lesions from osteoarthritis knees are characterized by sclerotic bone that is less well mineralized. Arthritis Res Ther. 2009;11(1):R11. doi: 10.1186/ar2601. Epub 2009 Jan 26. PMID 19171047
- See also: New England Baptist Hospital Website — http://www.nebh.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 4 orthopedic surgeons at one hospital between the dates of March, 2009 and April, 2013.
Groups:
- Enrolled: Inclusion Criteria:
  - subjects having primary knee replacement surgery
  Exclusion Criteria:
  * having a revision knee replacement instead of a primary knee replacement
  * contraindicated for MRI or CT scans
  * allergy to the contrast agent gadolinium
  * pregnant women
Period: Overall Study
Arm/Group | Enrolled
Started | 101
Completed | 60
Not Completed | 41
Not completed — unable/unwilling to complete MRI | 13
Not completed — specimen missed due to scheduling error | 14
Not completed — specimen unusable | 7
Not completed — Withdrawal by Subject | 3
Not completed — radiology error | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Groups:
- Enrolled: Subjects having primary knee replacement surgery
  Exclusion Criteria:
  * having a revision knee replacement instead of a primary knee replacement
  * contraindicated for MRI or CT scans
  * allergy to the contrast agent gadolinium
  * pregnant women
Arm/Group | Enrolled
Number analyzed (Participants) | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 55
  >=65 years | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.89 (8.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 51
Region of Enrollment [Number; unit: participants]
  United States | 101

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Viable Specimens for Genetic Analysis
Time Frame: Tissue samples collected at time of surgery
Measure: Number; unit: participants
Groups:
- Specimens: Viable specimens for genetic analysis
Arm/Group | Specimens
Number analyzed (Participants) | 60
participants | 14

ADVERSE EVENTS:
Groups:
- Enrolled: subjects having primary knee replacement surgery
Arm/Group | Enrolled
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No